CLINICAL TRIAL: NCT04109443
Title: Influences on Risk Behaviors Among Young Men
Brief Title: Young Men and Media Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-39323; K23MH109346 (NIH)
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Sexual Behavior
Keywords: Adolescent sexual minority males (ASMM); gay, bisexual, and other men who have sex with me (GBMSM); Online sexual health media literacy intervention; HIV prevention; Healthy sexual behaviors
MeSH Terms: conditions — Sexual Behavior; Homosexuality; Bisexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young Men & Media Program group (Experimental): Participants randomized to the Young Men and Media Program group will have access to the online sexual health media literacy materials. They will also complete three assessments at baseline, post-intervention, and a 3 month follow-up.
  Interventions: Behavioral: Young Men & Media Program
- Control group (Active Comparator): Participants randomized to the control group will have access to available websites (such as by the CDC) that provide information about sexual health and preventing sexually transmitted infections including HIV. They will complete three assessments at baseline, post-intervention, and a 3 month follow-up.
  Interventions: Behavioral: Available websites on safe sex and preventing STIs

INTERVENTIONS:
Behavioral: Young Men & Media Program — The online sexual health media literacy website includes content about (1) male anatomy; (2) HIV/STI prevention; (3) overall sexual health; and (4) sexually explicit online media (SEOM) literacy.
  Arms: Young Men & Media Program group
Behavioral: Available websites on safe sex and preventing STIs — Available websites (such as by the CDC) that provide information about sexual health and preventing sexually transmitted infections (STIs) including HIV.
  Arms: Control group

SUMMARY:
Adolescent sexual minority males (ASMM) continue to account for a disproportionate number of HIV infections in the United States. Racial and ethnic minority populations are particularly affected. Increased HIV rates reflect sexual risk behaviors during early sexual experiences. Research suggests that initial sexual risk-taking occurs during adolescence among sexual minority males. Therefore, it is important for HIV prevention interventions to target adolescent sexual minority males. Targeting sexual minority males during adolescence will help them learn and establish healthy sexual behaviors early in their psychosexual development, which will have both immediate and long-term health benefits.To promote adolescent sexual minority males' critical examination of online media and decrease their sexual risk-taking, this study proposes an exploratory clinical trial to pilot test an online sexual health media literacy intervention that was developed during formative research for feasibility and acceptability. Overall, the proposed research has the potential to reach a wide audience of sexual minority males early in their sexual development, ultimately decreasing their sexual risk-taking and reducing the number of new HIV infections in this population.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as sexual minority
* Have intentionally accessed SEOM
* Have a valid personal email address
* Be a US resident
* Be new to the study

Exclusion Criteria:

* Are unwilling or unable to provide informed assent
* Are unable to understand and read English
* Do not have the appropriate device and necessary software to experience all the intervention content

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — cisgender
Enrollment: 154 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly M Nelson, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred online at the study website. Based on responses to the online screener survey, 422 potential participants were identified and 225 of them agreed to complete the baseline screening. 183 actually completed the baseline screening and of those 29 were determined ineligible leaving a final sample of 154 who were consented/enrolled in the study.
Period: Overall Study
Arm/Group | Young Men & Media Program Group | Control Group
Started | 77 | 77
Completed | 67 | 65
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Young Men & Media Program Group | Control Group | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 77 | 77 | 154
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 77 | 77 | 154
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 41 | 39 | 80
  Latino | 20 | 20 | 40
  Black/African American | 9 | 8 | 17
  Mixed Race/Other | 7 | 9 | 16
  Not provided | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 77 | 77 | 154

OUTCOME MEASURES:

1. Primary Outcome: Study Feasibility Based on the Overall Recruitment Rate
Description: The overall recruitment rate will be calculated by dividing the total number of participants enrolled (n=154) by the total number of eligible potential participants from the initial online screener (n=422).
Time Frame: approximately 4.5 months
Population: Based on responses to the online screener survey, 422 potential participants were identified and 225 of them agreed to complete the baseline screening. 183 actually completed the baseline screening and of those 29 were determined ineligible leaving a final sample of 154 who were consented/enrolled in the study.
Measure: Number; unit: overall recruitment rate
Units Other Than Participants: percent recruited
Groups:
- All Eligible Participants: Based on responses to the online screener survey, 422 potential participants were identified.
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 154
Number analyzed (percent recruited) | 422
overall recruitment rate | 36.5

2. Primary Outcome: Study Feasibility Based on Banner ad Click Through Rate for All Participants Combined
Description: The banner click through rate will be calculated as the proportion of banner ads that participants click each week and then averaged for an overall rate at the end of study completion.
Time Frame: approximately 4.5 months
Population: The number of clicks on the banner ads could not be obtained from the system and therefore could not be reported.
Units Other Than Participants: Clicks
Groups:
- Participants Who Clicked the Banner: Total number of clicks on the banner ads.
Arm/Group | Participants Who Clicked the Banner
Number analyzed (Participants) | 0
Number analyzed (Clicks) | 0

3. Primary Outcome: Feasibility of the Media Literacy Intervention Based on Time Spent on the Intervention
Description: The time spent on each piece of intervention content will be determined from their online use.
Time Frame: 90 minutes
Population: For some intervention content, like viewing images, the investigators were not able to capture reliably how long participants stayed on a page due to the various ways that they could leave that page. Therefore, this outcome could not be measured reliably and the data are not presented.
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Number and Percentage of Participants Who Complete All the Intervention Content
Description: The online intervention will track what intervention content is viewed and the rate of participants who complete of all content will be calculated.
Time Frame: 90 minutes
Population: Outcome measure is only applicable to the Young Men & Media Program group.
Measure: Count of Participants; unit: Participants
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 77 | 0
Participants | 38 | 0

5. Primary Outcome: Mean Participant Satisfaction of the Intervention Content Areas Based on a 5 Star Rating System
Description: Participants will be asked to rate each of the 9 content area using a 5-star rating system where 1 star is the lowest and 5 stars is the highest rating. A mean of all ratings will be calculated. The closer the mean is to 5.0, the higher the satisfaction with the content areas. Participants will also be given the option of providing written feedback on each piece of content as well.
Time Frame: 90 minutes
Population: Only collected for intervention (Young Men & Media Program) group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 77 | 0
units on a scale | 4.3 (0.8) |

6. Primary Outcome: Count and Percentage of Participants Who Are Retained Through All Assessments
Description: The percentage of participants who completed all assessments divided by the number of enrolled participants
Time Frame: approximately 4.5 months
Population: All participants were combined to obtain the overall retention percent and number for the study.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants in the Study: All 154 participants combined from the Young Men & Media group (N=77) and the control group (N=77).
Arm/Group | All Participants in the Study
Number analyzed (Participants) | 154
Participants | 126

7. Secondary Outcome: Number of Sexual Partners
Description: Participants will be asked information about the number of sex partners in the prior 3 months.
Time Frame: Baseline, 3 months
Population: Data collection for this project concurred with the initial months of the COVID-19 pandemic in the United States. Although sexual behavior data were collected, our data indicates that at baseline the COVID-19 pandemic had already substantially reduced participants sexual contacts because most participants were no longer seeking out or interacting with sexual partners in-person. Thus, the validity and meaningfulness of these data are unclear.
Measure: Mean (Standard Deviation); unit: number of partners
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 77 | 77
number of partners
  Baseline | 0.49 (0.07) | 0.40 (0.07)
  3 months | 0.26 (0.07) | 0.23 (0.06)

8. Secondary Outcome: Number of Condomless Sex Acts With Male Partners
Description: Participants will be asked information about the number of condomless sex acts with male partners in the prior 3 months.
Time Frame: Baseline, 3 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: number of condomless sex acts
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 77 | 7
number of condomless sex acts
  Baseline | 0.39 (0.15) | 0.27 (0.09)
  3 months | 0.05 (0.04) | 0.10 (0.07)

9. Secondary Outcome: Change in 6-item Condom Use and Attitudes Scale
Description: Self-reported agreement with statements about condom use. Each item is scored 0-4 (0=strongly disagree; 4=strongly agree), yielding a total score of 0-24 with higher scores indicating more agreement that condom use interferes with sexual intimacy.
Time Frame: Baseline, 3 weeks, 3 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 77 | 77
score on a scale
  Baseline | 4.5 (1.3) | 4.2 (1.6)
  3 weeks | 4.9 (1.2) | 4.5 (1.5)
  3 months | 4.6 (1.5) | 4.9 (1.2)

10. Secondary Outcome: Change in 8-item Sexually Explicit Online Media (SEOM) Literacy Scale
Description: Self-reported agreement with statements about SEOM. Each item is scored 0-4 (0=strongly disagree; 4=strongly agree), yielding a total score of 0-32 with higher scores indicating more agreement with less SEOM literacy.
Time Frame: Baseline, 3 weeks, 3 months
Population: This scale was developed for this study and shows only acceptable internal reliability (Chronbach's alpha = 0.71, 0.75, 0.69). Results should be interpreted with caution as they may be unreliable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 77 | 77
units on a scale
  baseline | 17.43 (0.42) | 17.43 (0.42)
  3 weeks | 16.01 (0.38) | 16.6 (0.46)
  3 months | 16.7 (0.40) | 17.3 (0.41)

11. Secondary Outcome: Change in 4-item SEOM Knowledge Scale
Description: Self-reported assessment of True/False statements about SEOM. Each item will be scored as 0-1 (0=incorrect, 1=correct), yielding a total score of 0-4 with higher scores indicating higher levels of knowledge.
Time Frame: Baseline, 3 weeks, 3 months
Population: This scale was developed for this study and shows unacceptable internal reliability (Chronbach's alpha = 0.41, 0.38, 0.49). Results should be interpreted with caution as they are likely unreliable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 77 | 77
units on a scale
  baseline | 2.35 (0.13) | 2.36 (0.11)
  3 weeks | 2.97 (0.10) | 2.35 (0.12)
  3 months | 2.64 (0.14) | 2.61 (0.13)

12. Secondary Outcome: Knowledge of HIV and STI Transmission and Prevention
Description: A 52-item sexual health knowledge scale will be used to assess HIV/STI knowledge. The scale presents self-reported assessment of True/False statements about HIV and STI transmission and prevention. Each item will be scored as 0-1 (0=incorrect; 1=correct), yielding a total score of 0-52 with higher scores indicating higher levels of HIV/STI knowledge.
Time Frame: Baseline, 3 weeks, 3 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Young Men & Media Program Group | Control Group
Number analyzed (Participants) | 77 | 77
Score on a scale
  Baseline | 22.3 (7.9) | 22.4 (7.9)
  3 Weeks | 27.2 (7.0) | 24.3 (8.4)
  3 Months | 26 (7.7) | 25.5 (8.5)

ADVERSE EVENTS:
Time Frame: approximately 4.5 months
Arm/Group | Young Men & Media Program Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

LIMITATIONS AND CAVEATS:
Data collection for this project concurred with the initial months of the COVID-19 pandemic in the United States. As such, it is possible that some of the outcomes changed independent of the intervention. Additionally, the SEOM measures (outcomes 10 and 11) were developed for this study and appear to have some potential issues with internal reliability. As such, they should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT04109443/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT04109443/ICF_000.pdf